CLINICAL TRIAL: NCT07028996
Title: Clinical Investigation Plan for Non-CE-marked Medical Device Without Marking Objective (Category 4.4) to Evaluate Tolerance, Use and Performance of a Urine Collection Device (PEASY), in Hospitalized Patients: First-in-man Pilot Study
Brief Title: Tolerance, Use and Performance of the PEASY Urine Collection Device in Hospitalized Patients
Acronym: TUPELO
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: IDIL
Record Dates: First submitted 2025-06-03; First posted 2025-06-19 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Urinary Incontinence; Medical Device Discomfort
Keywords: Urinary incontinence; Penile clamp; Urinary sheath
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Daily use of the PEASY urine collection device for 5 days — The PEASY device features a non-adhesive attachment system to the penis, unlike penile sheaths which are used for the same indications and whose attachment system is based on an adhesive system. Fixation of the PEASY device to the penis involves the use of a clamp on the foreskin. The clamp has a certain elasticity and has been developed to be atraumatic.
  The medical device comprises a glans cup which covers the urinary meatus. This cup therefore rests on the glans.
Other: Daily collection of patient feedback using a visual analog scale (0-100) — Daily collection of patient feedback using a visual analog scale (0-100) and any suggestions for improving the device during an open interview at the end of the test period.

SUMMARY:
At present, 3 types of urine collection device can be distinguished: absorbent devices (diaper-type), penile clamps and penile collection sheaths. Both pads and penile sheaths are used depending on the department concerned, the clinical context and user preferences. A 2023 survey at Nîmes University Hospital showed that penis sleeves have undesirable side effects like fixation problems and pain on removal, and care assistants reported penile irritation caused by the penis sleeve. Caregivers also reported difficulties when handling and using penis sleeves.

There is clearly a need for a better device.To overcome the disadvantages of penis covers, the PEASY project team at Nîmes University Hospital has developed a practical, non-invasive medical device for eliminating urine, positioned on the glans: the PEASY device. This device is held in place by a non-adhesive fastening system that involves the foreskin, to ensure leakage-free urine flow.

DETAILED DESCRIPTION:
The problem of urine collection arises not only in incontinent patients, but also in continent patients who are unable to collect urine "actively". At present, three types of urine collection device can be distinguished: absorbent devices (diaper-type), penile clamps and penile collection sheaths. In the hospital, both pads and penile sheaths are used according to the department concerned, the patient's clinical context and user preferences. For example, 30,000 penis covers were used in 10 departments at the CHU de Nîmes in 2022.

However, a survey carried out at the CHU de Nîmes in 2023 showed that penis sleeves have undesirable side effects: 67% of care assistants reported fixation problems and pain on removal; 52% of care assistants reported penile irritation following use of the penis sleeve.

The survey also showed that the use of penis sleeves is not without its drawbacks: 76% of caregivers reported difficulties when handling and using penis sleeves.

There is a clear need for a device that i) reduces the irritation associated with penis sleeves, ii) is easy to insert and remove, and iii) guarantees no leakage.

To overcome the disadvantages of penis covers, the PEASY project team at Nîmes University Hospital has developed a practical, non-invasive medical device for eliminating urine, which is positioned on the glans penis: the PEASY device. This device is held in place by a non-adhesive fastening system that involves the foreskin, to ensure leakage-free urine flow.

To date, the hospital disposes of have a pre-production device which has never been tested on humans under real-life conditions. Before going any further with its development, all questions relating to its tolerance, usability and expected performance need to be addressed.

This is the aim of this pilot study, the results of which will enable the investigators to improve the device with a view to obtaining a finished product, or to discontinue its development.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring non-invasive urine collection.
* Incontinent patient for whom the use of a penile pouch to control leakage has been suggested by the care team.
* Uncircumcised patient.
* Patient with no physical anomaly preventing complete unhooding (phimosis, micropenis, penile invagination, etc.).
* Patient with no apparent irritation or infection of the glans (mycosis, herpetic lesion, etc.).
* Patient is conscious and able to answer simple questions.
* Patient has given free and informed consent.
* Patient has signed the consent form.
* Patient affiliated or beneficiary of a health insurance plan.

Exclusion Criteria:

* Patient participating in another high-risk interventional study.
* Patient in an exclusion period determined by another study.
* Patient under court protection, guardianship or curatorship.
* Patient unable to give consent.
* Patient for whom it is impossible to give informed information.
* Circumcised patients.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — People with penises
Study Population: For the purposes of the study, 20 incontinent patients for whom the use of a penile pouch to control leakage has been suggested by the care team, will be recruited from the active file of patients hospitalized in the Geriatric Medicine department of the CHU de Nîmes.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-06-18 (Estimated); Primary Completion 2025-12-03 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Daily measurement (at each change) from the patient's point of view. Pain in the glans | Day 1
  Pain in the glans will be recorded on a 0-100 visual analog scale in which 0 = no pain and 100 = worst possible pain.
Daily measurement (at each change) from the patient's point of view. Pruritis/burning in glans or foreskin | Day 1
  Pruritus/burning in the glans or foreskin will be recorded on a 0-100 visual analog scale in which 0 = no pruritis/burning and 100 = worst possible pruritis/burning.
Daily measurement (at each change) from the patient's point of view. Sensation of discomfort | Day 1
  Sensation of discomfort will be recorded on a 0-100 visual analog scale in which 0 = no discomfort and 100 = worst possible discomfort.
Daily measurement (at each change) from the patient's point of view. Pain in the glans | Day 2
  Pain in the glans will be recorded on a 0-100 visual analog scale in which 0 = no pain and 100 = worst possible pain.
Daily measurement (at each change) from the patient's point of view. Pruritis/burning in the glans or foreskin | Day 2
  Pruritis/burning in the glans or foreskin will be recorded on a 0-100 visual analog scale in which 0 = no pruritis/burning and 100 = worst possible pruritis/burning.
Daily measurement (at each change) from the patient's point of view. Sensation of discomfort | Day 2
  Sensation of discomfort will be recorded on a 0-100 visual analog scale in which 0 = no discomfort and 100 = worst possible discomfort.
Daily measurement (at each change) from the patient's point of view. Pain in the glans | Day 3
  Pain in the glans will be recorded on a 0-100 visual analog scale in which 0 = no pain and 100 = worst possible pain.
Daily measurement (at each change) from the patient's point of view. Pruritis/burning in the glans or foreskin | Day 3
  Pruritis/burning in the glans or foreskin will be recorded on a 0-100 visual analog scale in which 0 = no pruritis/burning and 100 = worst possible pruritis/burning.
Daily measurement (at each change) from the patient's point of view. Sensation of discomfort | Day 3
  Sensation of discomfort will be recorded on a 0-100 visual analog scale in which 0 = no discomfort and 100 = worst possible discomfort.
Daily measurement (at each change) from the patient's point of view. Pain in the glans | Day 4
  Pain in the glans will be recorded on a 0-100 visual analog scale in which 0 = no pain and 100 = worst possible pain.
Daily measurement (at each change) from the patient's point of view. Pruritis/burning in the glans or foreskin | Day 4
  Pruritus/burning in the glans or foreskin will be recorded on a 0-100 visual analog scale in which 0 = no pruritis/burning and 100 = worst possible pruritis/burning.
Daily measurement (at each change) from the patient's point of view. Sensation of discomfort | Day 4
  Sensation of discomfort will be recorded on a 0-100 visual analog scale in which 0 = no discomfort and 100 = worst possible discomfort.
Daily measurement (at each change) from the patient's point of view. Pain in the glans | Day 5
  Pain in the glans will be recorded on a 0-100 visual analog scale in which 0 = no pain and 100 = worst possible pain.
Daily measurement (at each change) from the patient's point of view. Pruritis/burning in the glans or foreskin | Day 5
  Pruritus/burning in the glans or foreskin will be recorded on a 0-100 visual analog scale in which 0 = no pruritis/burning and 100 = worst possible pruritis/burning.
Daily measurement (at each change) from the patient's point of view. Sensation of discomfort | Day 5
  Sensation of discomfort will be recorded on a 0-100 visual analog scale in which 0 = no discomfort and 100 = worst possible discomfort.
Daily measurement rom the caregiver's point of view | Day 1
  The following information will be recorded: appearance of erythema on the glans: Yes/No; appearance of erythema on the prepuce: Yes/No; patient's sensation of pain at the time of insertion: Yes/No; patient's sensation of pain at the time of removal: Yes/No
Daily measurement rom the caregiver's point of view | Day 2
  The following information will be recorded: appearance of erythema on the glans: Yes/No; appearance of erythema on the prepuce: Yes/No; patient's sensation of pain at the time of insertion: Yes/No; patient's sensation of pain at the time of removal: Yes/No
Daily measurement rom the caregiver's point of view | Day 3
  The following information will be recorded: appearance of erythema on the glans: Yes/No; appearance of erythema on the prepuce: Yes/No; patient's sensation of pain at the time of insertion: Yes/No; patient's sensation of pain at the time of removal: Yes/No
Daily measurement rom the caregiver's point of view | Day 4
  The following information will be recorded: appearance of erythema on the glans: Yes/No; appearance of erythema on the prepuce: Yes/No; patient's sensation of pain at the time of insertion: Yes/No; patient's sensation of pain at the time of removal: Yes/No
Daily measurement rom the caregiver's point of view | Day 5
  The following information will be recorded: appearance of erythema on the glans: Yes/No; appearance of erythema on the prepuce: Yes/No; patient's sensation of pain at the time of insertion: Yes/No; patient's sensation of pain at the time of removal: Yes/No

SECONDARY OUTCOMES:
A. Performance of PEASY from the caregiver's point of view: Bladder weakness | Day 1
  YES/NO
A. Performance of PEASY from the caregiver's point of view: Bladder weakness | Day 2
  YES/NO
A. Performance of PEASY from the caregiver's point of view: Bladder weakness | Day 3
  YES/NO
A. Performance of PEASY from the caregiver's point of view: Bladder weakness | Day 4
  YES/NO
A. Performance of PEASY from the caregiver's point of view: Bladder weakness | Day 5
  YES/NO
B. Performance of PEASY from the caregiver's point of view: facility of application | Day 1
  Question to caregiver: "How would you rate the application of the PEASY device? Visual analog scale 0-10 in which 0 is "very difficult" and 10 is "very easy".
B. Performance of PEASY from the caregiver's point of view: facility of application | Day 2
  Question to caregiver: "How would you rate the application of the PEASY device? Visual analog scale 0-10 in which 0 is "very difficult" and 10 is "very easy".
B. Performance of PEASY from the caregiver's point of view: facility of application | Day 3
  Question to caregiver: "How would you rate the application of the PEASY device? Visual analog scale 0-10 in which 0 is "very difficult" and 10 is "very easy".
B. Performance of PEASY from the caregiver's point of view: facility of application | Day 4
  Question to caregiver: "How would you rate the application of the PEASY device? Visual analog scale 0-10 in which 0 is "very difficult" and 10 is "very easy".
B. Performance of PEASY from the caregiver's point of view: facility of application | Day 5
  Question to caregiver: "How would you rate the application of the PEASY device? Visual analog scale 0-10 in which 0 is "very difficult" and 10 is "very easy".
C. Performance of PEASY from the caregiver's point of view: facility of removal | Day 1
  Question to caregiver: "How would you rate the removal of the PEASY device? Visual analog scale 0-10 in which 0 is "very difficult" and 10 is "very easy".
C. Performance of PEASY from the caregiver's point of view: facility of removal | Day 2
  Question to caregiver: "How would you rate the removal of the PEASY device? Visual analog scale 0-10 in which 0 is "very difficult" and 10 is "very easy".
C. Performance of PEASY from the caregiver's point of view: facility of removal | Day 3
  Question to caregiver: "How would you rate the removal of the PEASY device? Visual analog scale 0-10 in which 0 is "very difficult" and 10 is "very easy".
C. Performance of PEASY from the caregiver's point of view: facility of removal | Day 4
  Question to caregiver: "How would you rate the removal of the PEASY device? Visual analog scale 0-10 in which 0 is "very difficult" and 10 is "very easy".
C. Performance of PEASY from the caregiver's point of view: facility of removal | Day 5
  Question to caregiver: "How would you rate the removal of the PEASY device? Visual analog scale 0-10 in which 0 is "very difficult" and 10 is "very easy".
D- Evaluation by the caregiver of the the time required for the complete procedure (insertion and removal) of the PEASY device. Measured randomly by the Clinical Research Assistant. | Random measurements over 5 days
  Time required to insert the device: from decapping to connection of the PEASY to the urine collection bag tubing. Time required to remove the device. Total times in seconds
E.Qualitative evaluation by the caregiver of the various steps involved in applying the PEASY device | Day 5
  Questions to caregiver: "How do you rate each stage of using the PEASY device ? decapping, cup placement, recapping, PEASY device attachment, tubing connection. VAS 0-10 where 0 is "very difficult" and 10 is "very easy" for each step:
F. Usability of the PEASY device using the System Usability Scale questionnaire. | Day 5
  The system usability scale is a simple, ten-item attitude Likert scale giving a global view of subjective assessments of usability. Usability, as defined by the ISO standard ISO 9241 Part 11, can be measured only by taking into account the context of the system's use: i.e., who is using the system, what they are using it for, and the environment they are using it in. Measurements of usability have different aspects: effectiveness (can users successfully achieve their objectives) efficiency (how much effort and resources are expended to achieve those objectives) satisfaction (was the experience satisfactory). Measures of effectiveness and efficiency are context-specific. The System Usability Scale generally provides a high-level subjective view of usability and is often used to compare it between systems. It yields a single score on a scale of 0-100 in which 0 = completely unusable and 100 = extremely usable.
G. Success rate (%) of the PEASY | Day 5
  Success = the PEASY could be worn by the patient for 5 days. Description of the circumstances in the event of failure of the PEASY (device more in contact with the glans; device torn off; device under pressure with collection of urine at the foreskin; rejection by the patient; etc.).
  Success will be recorded as YES/NO: success = PEASY could be worn by patient for 5 days. Failure = use of penile sleeve and description of circumstances in case of failure.
H. User satisfaction from patient's point of view | Day 5
  User satisfaction with the PEASY device evaluated according to a visual analog scale of 0-100 in which 0 = completely dissatisfied and 100 = extremely satisfied.
H. User satisfaction from the caregiver's point of view | Day 5
  User satisfaction with the PEASY device evaluated according to a visual analog scale of 0-100 in which 0 = completely dissatisfied and 100 = extremely satisfied.
H. Suggestions for improving the PEASY device | Day 5
  Free collection of suggestions for improving the device by the patient and caregiver during an interview with the hospital CRA.
Summative evaluation of fitness for use according to EN62366:2015 | Day 5
  I. Five randomly-selected volunteer caregivers will be questioned on Day 5 about the PEASY device's suitability for use, using a summative suitability-for-use assessment questionnaire in accordance with standard EN62366:2015.

IPD SHARING:
Plan to Share IPD: No